CLINICAL TRIAL: NCT05203640
Title: Acute Glycemic Effects of Resistance Exercise in Post-menopausal Women With Type 1 Diabetes
Brief Title: Effects of Resistance Exercise on Blood Glucose in Post-menopausal Women With Type 1 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00112972
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Type 1 Diabetes
Keywords: resistance exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (Experimental): All participants will be in a single arm that undergoes two separate interventions. These interventions will include a high repetition, low resistance protocol, and a moderate repetition, moderate intensity protocol.
  Interventions: Behavioral: High repetition (HI); Behavioral: Moderate repetition (MOD)

INTERVENTIONS:
Behavioral: High repetition (HI) — Participants will perform 15 to 20 repetitions of 7 different exercises at 50% of their one repetition maximum
Behavioral: Moderate repetition (MOD) — Participants will perform 8 to 10 repetitions of 7 different exercise at 75-80% of their one repetition maximum

SUMMARY:
Regular physical activity has substantial health benefits in people with type 1 diabetes. The fear of hypoglycemia, both during and after exercise, is a major barrier to exercise in this population. A major obstacle to providing specific physical activity and exercise advice is that there are still significant gaps in the fundamental understanding of the impact of physical activity and exercise on blood glucose levels in type 1 diabetes.

Women with type 1 diabetes have a substantial increase in cardiovascular risk once they have passed menopause. They may lose both bone quality and muscle mass at a faster rate with aging than those without diabetes. Overall, these changes greatly increase the risk of both cardiovascular and frailty related complications. Despite the many potential benefits of resistance exercise for post-menopausal women with type 1 diabetes, there are currently no published studies examining the effects of resistance exercise in this population. Before being able to design a clinical trial of resistance exercise, an examination of the acute effects of resistance exercise on blood glucose levels in post-menopausal women with type 1 diabetes is required.

The present study will compare the glycemic effects of a low resistance, high repetition (3 sets of 15 to 20 repetitions) weight lifting program to the effects of a moderate resistance, moderate repetition (3 sets of 8 to 10 repetitions). The investigators hypothesize that the high repetition program will be associated with a bigger decline in blood glucose during exercise, but that the moderate resistance program will be associated with a higher risk of post-exercise hypoglycemia.

DETAILED DESCRIPTION:
Regular physical activity (PA) has substantial health benefits in people with type 1 diabetes (T1D). The fear of hypoglycemia, both during and after exercise, is a major barrier to exercise in this population. A major obstacle to providing specific PA advice is that there are still significant gaps in the fundamental understanding of the impact of PA and exercise on blood glucose levels in type 1 diabetes. For example, many of the existing studies were performed either uniquely with male participants, or with very few female participants. In addition to knowing little about the blood glucose response to PA and exercise in females with type 1 diabetes in general, less is known about how menopause and the hormonal changes and impacts of age affect these outcomes.

Women with T1D have a substantial increase in cardiovascular risk once they have passed menopause. In addition to this increased risk for cardiovascular disease (CVD), individuals with T1D may lose both bone quality and muscle mass at a faster rate with aging than those without diabetes. Overall, these changes greatly increase the risk of both cardiovascular and frailty related complications in females with T1D. Despite the many potential benefits of resistance exercise for post-menopausal females with T1D, there are currently no published studies examining the effects of resistance exercise in this population. There are, in fact, no published exercise interventions of any type of exercise in post-menopausal females with T1D. As such, current guidelines for insulin adjustment and carbohydrate intake around PA and exercise may be inappropriate for post-menopausal women with T1D.

Pre-test measures: Interested participants will be invited to the Physical Activity and Diabetes Laboratory on the main campus of the University of Alberta. Participants will be asked questions related to menopause, PA levels, and medication. Blood pressure and heart rate will also be measured. Where participants are eligible, anthropometric characteristics will be measured using standard protocols. A blood sample will be drawn for assessment of HbA1c. Those who meet all eligibility criteria and complete informed consent forms will be asked to complete the initial exercise tests. Participants will perform a submaximal aerobic capacity test. Indirect calorimetry will be used to assess oxygen consumption and carbon dioxide production and will be used to extrapolate the participant's aerobic capacity. Participants will then undergo a strength test for each of the seven exercises involved in the study, in order to estimate the their one repetition maximum (1RM - the maximum weight that can be lifted safely and with good form).

Testing sessions: Participants will be asked to arrive at the lab at around 4:00 pm for both sessions, which will be randomly assigned by tossing a fair coin. During the sessions, participants will be asked to perform a total of 7 resistance exercises (leg press, chest press, leg curls, lat pulldowns, seated row, shoulder press, and abdominal crunches). One trial will consist of 3 sets of 15 to 20 repetitions at 50-60% of the participants pre-determined 1RM, and the other will be 3 sets of 8 to 10 repetitions at 75-80% 1RM. Blood samples will be drawn at baseline, at the end of exercise, and an hour post-exercise via an IV catheter. Participants will be asked to match their daily food and insulin intake as closely as possible from one testing session to the next for the day before, day of and day after the testing session. Participants will be provided with log sheets to assist in this task and will also be asked to avoid strenuous exercise and alcohol intake.

A CGM sensor will be subcutaneously inserted by one of the investigators (trained by a group from the CGM manufacturer) into the anterior abdominal area of the participant approximately 3 days prior to the first testing session. The Dexcom G6 CGM will store glucose data every 5 minutes for up to 10 days. The participant will be instructed on how to remove their sensor at least 24 hours after the exercise session, and will be asked to upload their data to Dexcom Clarity to share with the study team. Background physical activity will be tracked using accelerometers.

Focus group/Interviews: After the exercise sessions have been completed, study participants will be invited to participate in a focus-group asking questions about their exercise experience, preferences between protocols, barriers to exercise, and other information they feel may improve their exercise experience. These focus groups will be conducted by a trained facilitator, and should take no more than two hours. For those who cannot attend the focus group, a video-conference to answer the questions in an interview format may be scheduled if they still wish to participate in this portion of the study.

ELIGIBILITY:
Inclusion Criteria:

* female
* type 1 diabetes diagnosed for at least 1 year
* at least 12 months since last menstrual period
* physically able and willing to perform resistance exercise
* HbA1c < 10%
* residing near Edmonton, Alberta / able to attend laboratory based sessions at the University of Alberta

Exclusion Criteria:

* Individuals with HbA1c >9.9%
* Frequent and unpredictable hypoglycaemia
* A change in insulin management strategy within two months of the study
* Blood pressure > 144/95,
* Severe peripheral neuropathy,
* A history of cardiovascular disease
* Musculoskeletal injuries affecting the ability to perform resistance exercise.
* Individuals who are treated with medications (other than insulin) that affect glucose metabolism (e.g. atypical antipsychotics, corticosteroids)
* A body mass index >30kg/m2,
* Smoking
* Moderate to high alcohol intake (>2 drinks per day)

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Blood glucose | from 0 minutes to 45 minutes, and from 45 minutes to 105 minutes
  Change in blood glucose during and after exercise

SECONDARY OUTCOMES:
Mean continuous glucose monitoring (CGM) glucose | 0 to 6 hours post exercise, overnight post exercise (midnight to 6 am) and 24 hours post exercise
  Interstitial glucose as measured by CGM
coefficient of variation (CV) | 0 to 6 hours post exercise, overnight post exercise (midnight to 6 am) and 24 hours post exercise
  CV of CGM glucose
standard deviation (SD) | 0 to 6 hours post exercise, overnight post exercise (midnight to 6 am) and 24 hours post exercise
  SD of CGM glucose
frequency of hypoglycemia | 0 to 6 hours post exercise, overnight post exercise (midnight to 6 am) and 24 hours post exercise
  number of times that CGM glucose was equal to or less than 3.9 mmol/L
frequency of hyperglycemia | 0 to 6 hours post exercise, overnight post exercise (midnight to 6 am) and 24 hours post exercise
  number of times that CGM glucose was equal to or above 10.0 mmol/L
percent time in range | 0 to 6 hours post exercise, overnight post exercise (midnight to 6 am) and 24 hours post exercise
  percentage of time spent between 4.0 and 9.9 mmol/L
percent time in hypoglycemia | 0 to 6 hours post exercise, overnight post exercise (midnight to 6 am) and 24 hours post exercise
  percentage of time spent equal to or below 3.9 mmol/L
percent time in hyperglycemia | 0 to 6 hours post exercise, overnight post exercise (midnight to 6 am) and 24 hours post exercise
  percentage of time spent at or above 10.0 mmol/L
carbohydrate supplementation | 0 to 45 minutes (during exercise)
  grams of carbohydrate provided to prevent hypoglycemia during exercise

CONTACTS AND LOCATIONS:
Locations (1):
- Alberta Diabetes Institute, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No